CLINICAL TRIAL: NCT05385900
Title: An Exploratory Study of Pembrolizumab Combined With Anlotinib and Chemotherapy Neoadjuvant Therapy of Locally Advanced Gastric Cancer
Brief Title: Immune Combined Targeted and Chemotherapy in Perioperative Treatment of Locally Advanced Gastric Cancer
Acronym: ICTCPTLAGC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQXB-GC-II-002
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — anlotinib; Drug Therapy; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Penpulimab in combination with anlotinib and chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab in combination with anlotinib and chemotherapy (Experimental): After receiving the corresponding neoadjuvant therapy for 3 cycles according to the established treatment plan, surgery should be performed within 3-6 weeks after drug withdrawal.
  Interventions: Drug: Penpulimab combination with anlotinib and chemotherapy

INTERVENTIONS:
Drug: Penpulimab combination with anlotinib and chemotherapy — Penpulimab: fixed dose of 200 mg, administered on day 1 of each cycle, repeated every 3 weeks; Anlotinib: 12 mg, administered on days 1-14 of each cycle, orally once a day, about half an hour before breakfast (the time of daily administration should be the same as possible), with warm water, every 3 weeks Repeat 1 time
  Other Names: Teggio; Oxaliplatin

SUMMARY:
An exploratory study of pembrolizumab combined with anlotinib and chemotherapy in the perioperative treatment of locally advanced gastric cancer

DETAILED DESCRIPTION:
Previous studies have shown that anti-vascular drugs have excellent anti-tumor effects in the neoadjuvant treatment of locally advanced gastric cancer. The purpose of this study was to evaluate the neoadjuvant treatment of locally advanced gastric cancer with Penpulimab combined with anlotinib and chemotherapy. pathological complete response rate, disease-free survival, objective response rate, R0 resection rate and safety. The subjects used in the study were patients with resectable or potentially resectable T3~4N+M0 gastric cancer who were confirmed by endoscopic ultrasonography and enhanced CT. The specific dosing schedule of Piamprimab combined with anlotinib and chemotherapy was adopted. After receiving the corresponding neoadjuvant therapy for 3 cycles, surgery should be performed within 3-6 weeks after drug withdrawal; it is recommended that patients be given corresponding Adjuvant therapy, the specific adjuvant therapy plan shall be formulated by the investigator according to the individual situation of the patient. The primary endpoint was pathological complete response rate, and secondary key indicators were disease-free survival, objective response rate, R0 resection rate, and safety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 70 years old, male or female;
* ECOG score 0~1 points;
* Patients with locally advanced gastric cancer (according to WHO 2015 classification) confirmed by pathology (histology or cytology);
* According to the eighth edition of clinical tumor TNM staging, patients with T3~4N+M0 gastric cancer confirmed by endoscopic ultrasonography and enhanced CT examination as resectable or potentially resectable;
* With measurable lesions (according to RECIST 1.1 criteria, the long diameter of CT scan of tumor lesions is ≥10mm, and the short diameter of CT scan of lymph node lesions is ≥15mm;), tumor diameter > 2cm;
* Those who were diagnosed with gastric cancer for the first time before enrolling in the group and who have not undergone radiotherapy, chemotherapy, surgery and targeted therapy;

  1. Major organ function is normal, that is, the following criteria are met:
  2. Routine blood tests must meet (no blood transfusion, no hematopoietic factor and no drug correction within 14 days):

     1. ANC ≥ 1.5×109/L；
     2. PLT ≥ 100×109/L；
     3. HB ≥ 90 g/L；
  3. Biochemical tests must meet the following criteria:

     1. TBIL≤1.5×ULN；
     2. ALT、AST≤ 2.5×ULN
     3. serum creatinines Cr≤1.5×ULN，endogenous creatinine clearance≥50 mL/min（Cockcroft-Gault formula）；
* Coagulation function must meet the following criteria：INR≤1.5×ULN;APTT≤1.5×ULN； Patients with myocardial ischemia or myocardial infarction above grade 1, arrhythmia (including QTc≥450ms (male), QTc≥470ms (female)) and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification);
* Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days before starting the study drug, and be willing to use a medically-approved high-efficiency contraceptive during the study and within 3 months after the last dose of study drug ( Such as: intrauterine device, contraceptive pill or condom); for male subjects whose partner is a female of childbearing age, surgical sterilization, or agree to use an effective method during the study and within 3 months after the last study dose contraception;
* The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up;

Exclusion Criteria:

* Target disease exclusion criteria

  1. Patients with distant metastasis;
  2. Subjects who have previously received anti-PD-1 (L1) or CTLA4 monoclonal antibody therapy;
* Medical history and comorbidities

  1. Suffering from other malignant tumors in the past 3 years;
  2. Suffering from any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, Hypothyroidism (may be included after hormone replacement therapy); patients with vitiligo or complete remission of childhood asthma who do not require any intervention in adulthood may be included; patients requiring medical intervention with bronchodilators are not included;
  3. The use of immunosuppressive drugs within 14 days before the first use of the study drug, excluding nasal and inhaled corticosteroids or systemic steroids at physiological doses (ie, no more than 10 mg/day prednisone or its equivalent) );
  4. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg despite optimal medical therapy);
  5. Patients with newly diagnosed angina pectoris within 3 months before screening or myocardial infarction events within 6 months before screening; arrhythmia (including QTcF: ≥450 ms for males, ≥470 ms for females) requires long-term use of antiarrhythmic drugs and New York Cardiac Association classification ≥ class II cardiac insufficiency; or uncontrolled heart failure;
  6. There is evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, and severely impaired lung function;
  7. Complicated severe infection within 4 weeks before the first dose (eg: need for intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever >38.5°C during the screening period/before the first dose;
  8. Clinically significant hemoptysis (more than 50 mL of hemoptysis per day) within 3 months before the study, or clinically significant bleeding symptoms or obvious bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic Gastric ulcer, fecal occult blood++ or above baseline, or suffering from vasculitis, etc.).
  9. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
  10. Administer live attenuated vaccines within 4 weeks before the first dose or during the study period;
* Physical examination and laboratory findings

  1. Patients with congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (positive hepatitis C antibody, and high HCV-RNA) (the lower limit of detection of the analytical method) or co-infection with hepatitis B and C;
  2. Pregnant or breastfeeding women; patients with childbearing potential who are unwilling or unable to take effective contraceptive measures;
  3. Known positive history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Allergies, anaphylaxis and adverse drug reactions

  1. Severe allergic reactions to other monoclonal antibodies;
  2. Allergy or intolerance to infusion;
  3. Have a history of severe allergy to Anlotinib or its preventive medicines;
* Subjects who are participating in other clinical studies or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or 5 half-lives of the research drug;
* The subject is known to have a history of psychotropic substance abuse, alcohol or drug abuse;
* The investigator believes that there are any conditions that may harm the subject or prevent the subject from meeting or performing the research requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response, pCR | 12months
  Defined as tumor tissue specimens resected surgically after neoadjuvant therapy with no residual tumor cells.

SECONDARY OUTCOMES:
major pathologic response, MPR | 12months
  Defined as tumor specimens resected after neoadjuvant therapy with residual tumor cells ≤10%

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hong, Study Chair — Air Force Military Medical University, China

IPD SHARING:
Plan to Share IPD: No